CLINICAL TRIAL: NCT00707252
Title: Phase I/II Study of Polyphenon E in Addition to Erlotinib in Advanced Non Small Cell Lung Cancer
Brief Title: Study of Polyphenon E in Addition to Erlotinib in Advanced Non Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Phase II not initiated due to cancellation of supply of Poly E by collaborator.
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Collaborators: Polyphenon E International,Inc. (Industry)
Responsible Party: Principal Investigator, Glenn Mills, Professor of Medicine, Louisiana State University Health Sciences Center Shreveport
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H06-128
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-small cell lung cancer; Erlotinib; Polyphenon E; Tarceva; Advanced Non-small Cell Lung Cancer Stage IIIb or IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — polyphenon E; Tea; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase I/II (Experimental): Phase I: Polyphenon E + Erlotinib - Polyphenon E 200, 400 and 800 mg/day dose levels evaluated in a step-wise manner with Erlotinib 150 mg/day to establish Maximum Tolerated Dose (MTD) of Polyphenon E. Phase II consists of MTD of Polyphenon E established in Phase I, administered alone for two weeks and thereafter together with Erlotinib 150 mg/day.
  Interventions: Drug: Polyphenon E; Drug: Tarceva

INTERVENTIONS:
Drug: Polyphenon E — Patients will be assigned to 3 sequential cohorts of three different dose levels of Polyphenon E (providing 200, 400 and 800mg of Polyphenon E given once daily) in a step-wise manner.
  Other Names: "Polyphenon extract, Green Tea"
Drug: Tarceva — All patients will also receive Erlotinib 150mg po/day from Day 1.
  Other Names: (Erlotinib)

SUMMARY:
The purpose of this study is to study if the addition of the green tea extract, Polyphenon E, to Erlotinib is safe and if it has potential to improve outcomes in second line therapy for Advanced Stage IIIb/IV Non-small cell lung cancer.

DETAILED DESCRIPTION:
To evaluate the short term effects of Polyphenon E administered alone and in combination with erlotinib to patients with advanced Stage IIIB or IV Non Small Cell Lung Cancer (NSCLC) that has progressed after first line chemotherapy. We will do a Phase I dose escalation study with Polyphenon E and a fixed dose of erlotinib to evaluate for any significant adverse events related to the combination.

Once the maximum tolerated dose (MTD) of Polyphenon E has been established the Phase II trial will be embarked upon using this dose in combination with erlotinib. In both the Phase I and Phase II parts the agents will administered until time of progression or unacceptable side effects occur.

The primary end point of the Phase I part is establishing the safety, tolerability and MTD of Polyphenon E in combination with erlotinib given at 150mg per day.

The Primary endpoint of the Phase II part that will be studied is Response rate (RR) to the combination. Progression free survival (PFS), Overall Survival (OS) and the safety and tolerability of Polyphenon E in addition to erlotinib in this subject population and setting will be assessed as secondary objectives.

Changes in serum markers related to progression of cancer will also be studied as part of the Phase I and phase II study. The effect of Polyphenon E with or without erlotinib on the serum levels of circulating c-met RNA, Interleukin-8 (Il-8), Hepatocyte Growth Factor (HGF) and Vascular Endothelial Growth Factor (VEGF) will be studied as secondary objectives. Epidermal Growth Factor Receptor (EGFR) expression of the initial tumor tissue and testing for EGFR mutations in the tumor tissue and serum DNA and evaluation of "KIRSTEN RAT SARCOMA VIRAL ONCOGENE HOMOLOG" (KRAS) mutations with correlation of these results with treatment outcome will also be undertaken as secondary objectives in both the Phase I and II parts.

1.1 Determine the safety, tolerability and MTD of Polyphenon E given in combination with erlotinib. Polyphenon E dose-escalation from 200, 400 and 800mg/day will be performed to evaluate for the MTD when used together with erlotinib 150mg/d.

1.2 Determine the effects of Polyphenon E in addition to erlotinib on response rate, progression free survival and overall survival

1.3 Determine the effects of Polyphenon E on circulating serum C-met messenger RNA

1.4 Determine the effects of Polyphenon E on serum HGF levels

1.5 Determine the effects of Polyphenon E on serum Il-8 levels

1.6 Determine the effects of Polyphenon E on serum VEGF levels 1.7 Determine the safety and tolerability of Polyphenon E in addition to erlotinib in this subject population

1.8 Determine the possible correlation between EGFR expression on original tumor tissue, EGFR mutations in tumor tissue and serum DNA and the presence of KRAS mutations with the treatment response and outcome.

This study was intended to be a Phase I/II study. This study never moved into the Phase II portion of the study. The sponsor stopped supplying Polyphenon E and there was not enough of a supply in-house to continue with Phase II.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven NSCLC
2. Stage IIIB or IV measurable disease burden after routine staging work up.
3. Documented disease progression after first or second line chemotherapy. This will be assessed using the Response Evaluation Criteria in Solid Tumors (RECIST)
4. Ability to give informed consent and willingness to adhere to study protocol
5. Ability to take oral medication
6. Age ≥ 18 years.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status between 0-2
8. Adequate hematological, hepatic and renal function defined as below:

   granulocyte count > 1500/mm3, platelet count > 100.000/mm3, serum creatinine < 1.5; bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase (ALP) at or below institutional upper limit of normal (IULN). All lab values should be obtained within 14 days of registration.
9. Patients have to have recovered from any toxic effects of prior chemotherapy or radiation therapy to a Grade 1 or less (except from alopecia). Enrollment should occur no less than 28 days after completion of prior therapy.
10. Ability to comply with the use of contraceptive measures starting 1 week before and ending 2 weeks after the last dose of study drug.

Exclusion Criteria:

1. Liver or kidney problems that would interfere with metabolism of study drug. This includes any preexisting elevation of AST, ALT, ALP or bilirubin.
2. Any condition that would hamper informed consent or ability to comply with the study protocol
3. Participation in another research study in the last three months
4. Known malignancy at any site other than NSCLC
5. Recent consumption of green tea (5 or more cups per day within one week of study enrollment)
6. Significant history of cardiac disease, e.g. uncontrolled hypertension, unstable angina, congestive-heart failure, myocardial infarction within the last six months or ventricular arrhythmias requiring medication.
7. Presence of metastatic brain lesions
8. Documented history of bleeding diathesis
9. Need to be on therapeutic anticoagulation
10. Pregnant and lactating women
11. Patients with a known seizure disorder who are taking Phenytoin, Carbamazepine or Phenobarbital
12. Patients taking medications known to interfere with erlotinib metabolism as listed below.

    * Atazanavir
    * Clarithromycin
    * Indinavir
    * Itraconazole
    * Ketoconazole
    * Nefazodone
    * Nelfinavir
    * Ritonavir
    * Saquinavir
    * Telithromycin
    * Troleandomycin
    * Voriconazole
    * Rifampicin
    * Rifabutin
    * Rifapentine
    * Phenytoin
    * Carbamazepine
    * Phenobarbital
    * St John's Wort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Phase 1: Number of Participants with Adverse Events. | At Screening and every week for first 4 weeks and then week 6, 8 and then every 4 weeks in Phase I study. Liver function tests will be monitored at least every 4 weeks as applicable. The patients will be followed up to 2 years on average.
  Toxicity evaluation of all adverse events monitored by physical exam, weight, vital signs, Complete Blood Count (CBC), Complete Metabolic Panel (CMP), coagulation panel and Computed Tomography (CT) scans of the chest, abdomen and pelvis, CT/Magnetic Resonance Imaging (MRI) of the head.
Phase 1: Maximum Tolerated Dose | Day 1 of Phase I until progression, death or intolerable side effects would occur. The patients will be followed up to 2 years on average.
  Dose-Limiting Toxicity (DLT) is defined as two or more events with grade 3 toxicity or a single event with grade 4-5 toxicity possibly or probably related to the study medications at a specific dose of Polyphenon E.
Phase 2: Response Rate | Start of Phase 2 to until progression, death or intolerable side effects occur. The patients will be followed up to 2 years on average.
  Response Rate defined as Complete (CR) + Partial Response (PR) using RECIST criteria.
  Complete response (CR):
  Complete disappearance of all measurable and non-measurable disease, no new lesions, no disease related symptoms, and normalization of markers and other abnormal lab values. All disease must be assessed using the same technique as baseline.
  Partial Response (PR):
  Applies only to patients with at least one measurable lesion. Greater than or equal to 30% decrease under baseline of the sum of longest diameters of all target measurable lesions. No unequivocal progression of non measurable disease. No new lesions. All target measurable lesions must be assessed using the same techniques as baseline.

SECONDARY OUTCOMES:
Phase I: Response rate | From registration until progression or intolerable side effects occur. The patients will be followed up to 2 years on average.
  Response Rate defined as Complete (CR) + Partial Response (PR) using RECIST criteria.
  Complete response (CR):
  Complete disappearance of all measurable and non-measurable disease, no new lesions, no disease related symptoms, and normalization of markers and other abnormal lab values. All disease must be assessed using the same technique as baseline.
  Partial Response (PR):
  Applies only to patients with at least one measurable lesion. Greater than or equal to 30% decrease under baseline of the sum of longest diameters of all target measurable lesions. No unequivocal progression of non measurable disease. No new lesions. All target measurable lesions must be assessed using the same techniques as baseline.
Phase 1: Progression Free Survival | From registration until progression or intolerable side effects occur. The patients will be followed up to 2 years on average.
  Progression- Free Survival:
  From date of registration to date of first observation of progressive disease, death due to any cause or symptomatic deterioration.
Phase 2: Progression Free Survival | From registration until progression or intolerable side effects occur. The patients will be followed up to 2 years on average.
  From date of registration to date of first observation of progressive disease, death due to any cause or symptomatic deterioration.
Phase 2: Overall Survival | From registration until progression or intolerable side effects occur. The patients will be followed up to 2 years on average.
  Time from registration to death of any cause measured in months.
Phase 2: Correlation between level of EGFR expression on the original tumor tissue and the presence of EGFR mutations in exons 18, 19 and 21 in serum DNA and original tumor tissue with the treatment response and outcome. | Pre-study until progression or intolerable side effects occur. The patients will be followed up to 2 years on average.
  To analyze signaling pathway activity western blot analysis will be performed using antibodies that recognize serum interleukin-8 (IL-8), VEGF and HGF levels. The level of circulating C-met RNA will be measured using Real Time Polymerase Chain Reaction (RT-PCR).
Phase 2: Correlation of KRAS mutations (in exons 2 and 3) in the original tumor tissue with treatment response and outcome. | Pre-study until progression or intolerable side effects occur. The patients will be followed up to 2 years on average.
  Clinical assay for detecting mutations in KRAS (direct sequencing).

CONTACTS AND LOCATIONS:
Overall Officials: Glenn M Mills, MD, Principal Investigator — LSU Health Sciences Center - Shreveport
Locations (1):
- LSUHSC-Shreveport, Feist-Weiller Cancer Center, Shreveport, Louisiana, United States